CLINICAL TRIAL: NCT02165072
Title: Inferior Vena Cava Collapsibility Index in Patients With Acute Kidney Injury
Brief Title: Inferior Vena cavaCollapsibility Index in Patients With Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L14-052
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Acute Kidney Injury
Keywords: Inferior vena cava; Kidney injury; Ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study that will examine the possibility of determining the type of Acute Kidney Injury (AKI) using bedside ultrasound machines.

DETAILED DESCRIPTION:
The investigators hypothesize that different types of AKI (pre-renal, renal, and post-renal) are associated with different inferior vena cava diameters and collapsibility index. The investigators will include subjects ages 18-89 years with AKI (creatinine of 2mg/100ml or higher for less than 24 hours from baseline creatinine ≤1.2 or with unknown baseline creatinine). Standard of care treatment will not be different for patients taking part in this study. Participants will have bedside ultrasounds on days 0, 1, and 3, and baseline and follow-up data will be collected from medical records.

ELIGIBILITY:
Inclusion Criteria:

1. Creatinine of 1.7 mg/100ml or higher for less than 24 hours from baseline creatinine ≤1.2 or with unknown baseline creatinine
2. Age range: 18-89 years
3. Age range ≥ 18

Exclusion Criteria:

1. Only chronic renal disease will exclude a patient from our study regardless of past medical history and medications they are taking. (For the purposes of this study, any patient with creatinine higher than 1.2 mg /100ml for more than 24 hours will be identified as having chronic renal disease.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ages 18-89 years with AKI (creatinine of 1.7mg/100ml or higher for less than 24 hours from baseline creatinine ≤1.2 or with unknown baseline creatinine). Standard of care treatment will not be different for patients taking part in this study. Participants will have bedside ultrasounds on days 0, 1, and 3, and baseline and follow-up data will be collected from medical records.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Nugent, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech Univrsity Health Science Center, Lubbock, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound of Acute Kidney Injury: This study represents a convenience sample of patients admitted to a medical intensive care unit with laboratory evidence of acute kidney injury. This is a prospective study. There is one study group only. There is no randomization.
Period: Overall Study
Arm/Group | Ultrasound of Acute Kidney Injury
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound of Acute Kidney Injury
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum and Minimum Diameters of the Inferior Vena Cava in Patients With Acute Kidney Injury
Description: The investigators will measure the maximum and minimum diameters of the inferior vena cava with patients with acute kidney injury.
Time Frame: Day 1 of ICU admission
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ultrasound of Acute Kidney Injury
Number analyzed (Participants) | 30
cm
  Maximum diameter | 1.8 (0.5)
  Minimum diameter | 1.2 (0.6)

2. Primary Outcome: Percent Collapse of the Inferior Vena Cava in Patients With Acute Kidney Injury
Description: The investigators will measure the maximum and minimum diameters of the inferior vena cava with patients with acute kidney injury and calculate the percent change between the maximum and minimum diameters.
Time Frame: Day 1 of ICU admission
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ultrasound of Acute Kidney Injury
Number analyzed (Participants) | 30
Percent change | 32 (20)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire study period of approximately 1 year.
Description: This study involved using abdominal ultrasound to measure the inferior vena cava dimensions. This required a short interaction with the patient making this routine measurement with a bedside ultrasound. There were no adverse events
Arm/Group | Ultrasound of Acute Kidney Injury
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
This study is straightforward and involves measurements of the inferior vena cava. The study population was heterogeneous. Study measurements depend on the ability to identify the inferior vena cava with precision and make accurate measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No